CLINICAL TRIAL: NCT02236780
Title: Influence of Environmental Conditions on In Vitro Fertilization (IVF) Attempts and Induced Pregnancies
Acronym: MeteoFIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: UPRES EA 2506 (Santé-Environnement-Vieillissement), France (Unknown)
Responsible Party: Sponsor
Other Study IDs: AOR13130
Record Dates: First submitted 2014-09-08; First posted 2014-09-11 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: In Vitro Fertilisation; Environmental Conditions
Keywords: in vitro fertilisation; environmental conditions; pregnancy; live birth rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main purpose of the study is to assess the impact of environmental conditions on live-birth rates after intraconjugal IVF.

The second purposes are

* to assess the impact on pregnancies (prematurity, preeclampsia);
* to assess the impact on newborn's health (stunted growth);
* to evaluate the consistency of results observed between assisted pregnancies and spontaneous pregnancies.

DETAILED DESCRIPTION:
This multicenter epidemiological study aims to analyze the individual standardized clinical records, collected prospectively since 2008 in the medically assisted procreation centers (MAP).

These individual data will be mapped to the environmental data (meteorological and air quality), recorded in the area of residence of the mother at the time of conception and pregnancy, as well as to the socio-economic data.

Choice of centers:

* The study will be proposed to the 106 private or public centers in metropolitan France who are authorized for MAP procedures such as IVF and ICSI.
* Only the centers who perform more than 200 oocyte retrievals per year will be selected to participate in the study.

More than 80% of attempts performed by the selected centers should be available (without missing data) on the induced pregnancies and their outcome (minimum data set for each case: age of man and woman, cause of infertility, technique used, sperm collection method (ejaculation, surgical sperm retrieval techniques), total number of embryos obtained, clinical pregnancy or not, term of pregnancy, weight and height of the child at birth).

ELIGIBILITY:
Inclusion Criteria:

* Intraconjugal IVF and ICSI
* Transfers of frozen embryos after intraconjugal IVF or ICSI

Exclusion Criteria:

* IVF and ICSI with sperm donation
* IVF and ICSI with egg donation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study focuses on intraconjugal IVF attempts (conventional IVF, microinjection intra-cytoplasmic sperm injection (ICSI) and frozen embryo transfers) realised for MAP procedures in metropolitan France, in the period of 01/01/2008 to 12/31/2012 (5 years).
Sampling Method: Non-Probability Sample
Enrollment: 24000 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 1 year
  Live birth rate after intraconjugal IVF (IVF and ICSI) by oocyte retrieval and by embryo transfer.

SECONDARY OUTCOMES:
Fertilization rate | 1 year
  Rate of fertilization (IVF and ICSI), rate of good quality embryos, rate of blastoformation (if prolonged culture), rate of embryo freezing.
Rates of clinical pregnancy | 1 year
  Rates of assisted pregnancy, rate of spontaneous miscarriage, rate of medical termination of pregnancy, rate of pathology of pregnancy (pre-eclampsia, gestational diabetes, placenta praevia, signs of preterm labor with hospitalization).
Fetal growth restriction rate | 1 year
  Fetal growth restriction rate, biometrics of child at birth (height, weight, head circumference, Body Mass Index), preterm birth rate, transfer rate to intensive care units.
Effect sizes and periods of susceptibility to environmental conditions | 5 years
  Effect sizes and periods of susceptibility to environmental conditions among assisted pregnancies and spontaneous pregnancies.

CONTACTS AND LOCATIONS:
Overall Officials: Alain BEAUCHET, MD, Study Chair — Hôpital Ambroise Paré, AP-HP; Philippe AEGERTER, MD, PhD, Study Director — Hôpital Ambroise Paré, AP-HP; Rachel LEVY, MD, PhD, Study Director — Hôpital Jean Verdier, AP-HP
Locations (1):
- Alain BEAUCHET, Boulogne-Billancourt, Hauts-de-seine, France